CLINICAL TRIAL: NCT02242838
Title: Post-Marketing Surveillance of Micardis® (Telmisartan) Special Drug Use-results Survey on Long-term Treatment
Brief Title: Post-Marketing Surveillance of Micardis® (Telmisartan) in Patients With Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.500
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hypertensive patients
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan
  Other Names: Micardis®

SUMMARY:
The primary objective of this survey is to prospectively investigate safety and efficacy in patients with hypertension treated with telmisartan in proper use in medical practice over a long period

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension

Exclusion Criteria:

Patients with the following conditions

* Patients with a history of hypersensitivity of this product
* Women in pregnancy (included the possibility of pregnancy)
* Patients with severe biliary obstructive disorders or severe hepatic insufficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hypertension patients without telmisartan treatment are selected at medical institutions
Sampling Method: Non-Probability Sample
Enrollment: 6336 (Actual)
Dates: Start 2003-09; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse drug reactions | up to 1 year
Incidence of adverse drug reactions | up to 1 year
  classified by Medical Dictionary for Regulatory Activities (MedDRA) terminology
Change in Mean systolic blood pressure (SBP) | up to 1 year
Change in Mean diastolic blood pressure (DBP) | up to 1 year

SECONDARY OUTCOMES:
Overall assessment of efficacy by investigator on 4-point scale | at 3 month, after 1 year
Change in pulse rate | up to 1 year